CLINICAL TRIAL: NCT00955214
Title: Impact of Paclitaxel-eluting Stent for Small Coronary Artery Disease
Brief Title: Small Coronary Artery Treated by TAXUS Liberté Registry in Japan
Acronym: SACRA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Society for Advancement of Coronary Intervention Research (Network)
Responsible Party: Kenya Nasu, Society for Advancement of Coronary Intervention Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SACRA1
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Stable Angina Pectoris; Unstable Angina Pectoris
Keywords: TAXUS Liberté; Small coronary artery disease; Paclitaxel-eluting stent
MeSH Terms: conditions — Angina, Stable; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2.5mm Paclitaxel-eluting stent (Experimental)
  Interventions: Device: TAXUS Liberté paclitaxel-eluting coronary stent system

INTERVENTIONS:
Device: TAXUS Liberté paclitaxel-eluting coronary stent system — diameter is 2.5mm

SUMMARY:
The utilization of paclitaxel-eluting coronary stents in small vessel diseases is effective in reducing both repeat revascularization and major adverse cardiac events within two year follow-up. To evaluate the procedural, short and long term clinical outcomes of the Taxus Liberte™ Paclitaxel-Eluting Coronary Stent in small coronary arteries of ≤ 2.5 mm in the reference vessel diameter.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years and are able to undergo CABG
2. Females who are not pregnant
3. Patients who present with angina symptoms or myocardial ischemia
4. Patients available for post-procedural observation and coronary angiography at 24 months
5. Patients who have signed patient informed consent
6. Lesion which is eligible for only one 2.5mm paclitaxel-eluting stent
7. De novo lesion or non-stented restenosed lesion

Exclusion Criteria:

1. Patients contraindicated for antiplatelet therapy or anticoagulant therapy
2. Patients with significant allergic reaction to contrast medium
3. Chronic total occlusion
4. Lesion with TIMI0
5. Lesion which is needed more than two stents
6. Patients with chronic renal failure (SCr>3.0mg/dl) -

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Target lesion revascularization rate | within 9months

SECONDARY OUTCOMES:
Technical success | initial
Target lesion revascularization rate | 12 months
Target lesion revascularization rate | 24 months
Target vessel revascularization rate | 12 months
Target vessel revascularization rate | 24 months
The rate of MACE including MI due to stent thrombosis | 12 months
The rate of MACE including MI due to stent thrombosis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenya Nasu, MD, Principal Investigator — Toyohashi Heart Center; Yuji Oikawa, MD, Principal Investigator — Cardiovascular institute hospital
Locations (23):
- Japan (23):
  - Japanese red cross nagoya daiichi hospital, Nagoya, Aichi-ken
  - Higashi Cardiovascular clinic, Toyohashi, Aichi-ken
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - Kokura memorial hospital, Kitakyushu, Fukuoka
  - Hoshi general hospital, Kōriyama, Fukushima
  - Southen tohoku research institute for neuroscience, Kōriyama, Fukushima
  - Gunma prefectural cardiovascular center, Maebashi, Gunma
  - Asahikawa medical college hospital, Asahikawa, Hokkaido
  - Hakodate central general hospital, Hakodate, Hokkaido
  - Shinko kakogawa hospital, Kakogawa, Hyōgo
  - Okamoto general hospital, Uji, Kyoto
  - Miyagi cardiovascular and respiratory center, Kurihara, Miyagi
  - Rinku general medical center, Izumiōtsu, Osaka
  - Sakurabashi watanabe hospital, Osaka, Osaka
  - Shuwa general hospital, Kasukabe, Saitama
  - Kasukabe chuo general hospital, Kasukabe, Saitama
  - Kusatsu Heart Center, Kusatsu, Shiga
  - Ayase heart hospital, Adachi City, Tokyo
  - The cardiovascular institute hospital, Minato, Tokyo
  - Tokyo metropolitan police hospital, Naka, Tokyo
  - JR tokyo general hospital, Shibuya City, Tokyo
  - Tokyo medical university hospital, Shinjuku, Tokyo
  - Itabashi Chuo medical center, tabashi City, Tokyo

REFERENCES:
- [Background] Turco MA, Ormiston JA, Popma JJ, Hall JJ, Mann T, Cannon LA, Webster MW, Mishkel GJ, O'Shaughnessy CD, McGarry TF, Mandinov L, Dawkins KD, Baim DS. Reduced risk of restenosis in small vessels and reduced risk of myocardial infarction in long lesions with the new thin-strut TAXUS Liberte stent: 1-year results from the TAXUS ATLAS program. JACC Cardiovasc Interv. 2008 Dec;1(6):699-709. doi: 10.1016/j.jcin.2008.09.007. PMID 19463387
- [Background] Ahmed WH. Review of the TAXUS Liberte SR paclitaxel-eluting coronary stent. Expert Rev Med Devices. 2007 Mar;4(2):117-20. doi: 10.1586/17434440.4.2.117. PMID 17359218
- [Background] Elezi S, Dibra A, Mehilli J, Pache J, Wessely R, Schomig A, Kastrati A. Vessel size and outcome after coronary drug-eluting stent placement: results from a large cohort of patients treated with sirolimus- or paclitaxel-eluting stents. J Am Coll Cardiol. 2006 Oct 3;48(7):1304-9. doi: 10.1016/j.jacc.2006.05.068. Epub 2006 Sep 12. PMID 17010786